CLINICAL TRIAL: NCT05076539
Title: A Quantitative Assessment of Early Mobility in Total Knee Replacement Patients Using Smart Activity Tracker
Acronym: Geospatial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Curtin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Geospatial; 2017-2972 (Other: Singhealth)
Record Dates: First submitted 2021-09-20; First posted 2021-10-13 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Geospatial (Other): 50 patients will be issued a Garmin GPS-activity tracker where they will be required to wear for 24 hours for 1 week, prior to each timepoint (pre-operatively and 6 months post surgery)
  Interventions: Other: Garmin GPS activity tracker

INTERVENTIONS:
Other: Garmin GPS activity tracker — 50 patients will be issued a Garmin GPS-activity tracker where they will be required to wear for 24 hours for 1 week, prior to each timepoint (pre-operatively and 6 months post surgery).

SUMMARY:
This study aims to evaluate the patients' mobility and quality of life prior to their total knee replacement surgery and their progress pre-operatively and 6 months post-operatively using the smart activity tracker. We hypothesize that mobility limitation presents a strong correlation with reduced quality of life.

DETAILED DESCRIPTION:
The present study is to determine the effect of TKA based on their mobility and QOL pre and post surgery. The GPS and accelerometry-based tracker will be able to provide quantitative-based outcomes to indicate the physical activity of patients after TKR remains at or above pre-surgical levels.

A total of 50 participants are to be enrolled in this cross-sectional study. Patients who will be required to undergo unilateral total knee replacement will be recruited when fulfilling the respective inclusion and exclusion criteria. The patients will undergo the standard consultations and rehabilitation pre - and post operative care, no changes to the treatment itself will be made. After recruitment and counseling by the surgeon for TKR, the patients will have pre-operative baseline clinical scores taken prior to surgery. They will subsequently have their TKR surgery. Post-operatively, they will be followed up prospectively at the clinics as well as Orthopaedics Diagnostic Centre. Their outcome will be evaluated using validated scoring system, Oxford Knee Score, SF-36, Knee Society Clinical Rating System, satisfaction questionnaire, as well as be provided with a GPS-activity tracker.

50 patients will be issued a Garmin GPS-activity tracker where they will be required to wear for 24 hours for 1 week, prior to each timepoint (pre-operatively and 6 months post surgery). The de-identified raw data gathered from the Garmin tracker will be collected by Curtin University for their analysis.

The patients will undergo the standard consultations and rehabilitation pre - and postoperative care, no changes to the treatment itself will be made.

Standard consultations/review by orthopaedic specialist

* Pre-surgery
* 6 months post surgery

Standard Orthopaedic Diagnostic Center (ODC) data collection timepoints

* Pre-surgrey
* 6 months

Standard rehabilitation care

* Upon discharge
* 2 - 3 weeks post discharge in outpatient services (OPS)

On top of the standard consultations and rehabilitation pre - and postoperative care, the patients will be monitored on their normal lifestyle at home using a tracker worn on their wrists for 1 week, pre-operatively and 6 months post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are referred by the Orthopaedic surgeon and are diagnosed with Knee Osteoarthritis, and consented to unilateral total knee replacement.
* Able to ambulate with or without walking aid.
* Ability to provide informed consent.

Exclusion Criteria:

* Patients who have severe bilateral Knee Osteoarthritis, affecting their ability to walk and only one will be operated on.
* Patients with pre-existing cognitive issues, such as dementia.
* Patients planning for another surgery within 6 months after their TKR.
* Patients with existing co-morbidities that limit their walking ability, such as severe respiratory distress syndromes.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-11 (Actual); Primary Completion 2022-10-13 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Knee Society Clinical Rating system | pre-surgery
  Measuring knee range of motion, knee extension lag, knee alignment in standing using the knee society clinical rating system (KSS Scores)
Knee Society Clinical Rating system | 6 months post surgery
  Measuring knee range of motion, knee extension lag, knee alignment in standing using the knee society clinical rating system (KSS Scores)
Oxford Knee | pre-surgery
  Using the Oxford Knee questionnaire to get the oxford knee score
Oxford Knee | 6 months post surgery
  Using the Oxford Knee questionnaire to get the oxford knee score
SF 36 Health survey | pre-surgery
  SF36 questionnaires to get SF-36 scores
SF 36 Health survey | 6 months post surgery
  SF36 questionnaires to get SF-36 scores
Expectation met for surgery | pre-surgery
  Patient satisfaction form
Expectation met for surgery | 6 months post surgery
  Patient satisfaction form
Overall result of surgery | pre-surgery
  Subject's summary and outcomes form; data collected from Orthopaedic diagnostis center (ODC)
Overall result of surgery | 6 months post surgery
  Subject's summary and outcomes form; data collected from Orthopaedic diagnostis center (ODC)
Length of stay | up to 6 months post surgery
  the number of nights spend in the hospital from the day of surgery
Premorbid history | up to 6 months post surgery
  Patients reported ambulation status before surgery, including the use of walking aids and assistance level required
Early ambulation rate | up to 6 months post surgery
  Percentage of patients who start walking postoperative day (POD) 1
Knee range-of-motion | up to 6 months post surgery
  measure knee ROM
Ability to perform a straight leg raise | up to 6 months post surgery
  If patient is able to lift their leg independently. Lag is measured by a goniometer measured by a goniometer
Type of walking aids used | up to 6 months post surgery
  The type of walking aids required, namely, walking frame, broad- and narrow-based quadstick, or walking stick (in descending order of base of support provided)
Discharge Destination | up to 6 months post surgery
  Where the patient will be going to after discharge from SGH
Data Collected from Garmin GPS-activity tracker | Pre-surgery for 1 week
  1. Latitude and longitudinal location coordinates to determine an individual's activity space
  2. Distance travelled
  3. Walking speed
  4. Heart rate
  5. Calories burned
  6. Energy expenditure
  7. Steps count
  8. Physical activity
Data Collected from Garmin GPS-activity tracker | 6 months post surgery for 1 week
  1. Latitude and longitudinal location coordinates to determine an individual's activity space
  2. Distance travelled
  3. Walking speed
  4. Heart rate
  5. Calories burned
  6. Energy expenditure
  7. Steps count
  8. Physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Celia Tan Ia Choo, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No